CLINICAL TRIAL: NCT06758050
Title: Effect of Adding Core Exercises to Hip and Knee-focused Exercises on Patellofemoral Pain Syndrome
Brief Title: Effect of Core Exercises on Patellofemoral Pain Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Rana Ibrahim, Rana Ibrahim Ahmed Mahmoud, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: No:P.T.REC/012/005347
Record Dates: First submitted 2024-12-26; First posted 2025-01-03 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2024-12

CONDITIONS: Patellofemoral Pain Syndrome
Keywords: core strengthening exercises, hip and knee-focused exercises, patellofemoral pain syndrome
MeSH Terms: conditions — Patellofemoral Pain Syndrome

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): Group B (study group) (core strengthening exercises added to evidence-based approaches group) The core muscle strength training program The core muscle strength training program will last for 6 weeks and comprise of two training sessions per week, with a total of 12 sessions for the study group.
  During the main part of the training, the "big 3" exercises as described by McGill will be conducted. These include the curl-up, side bridge, and quadruped position.
  Interventions: Other: Core strengthening exercises; Other: Traditional treatment
- Control group (Active Comparator): Group A (control group) (evidence-based approaches group): The participants in the control group will receive only a hip and knee- focused exercise program.
  1. Hip-focused exercise: Based on previous studies, hip-focused exercises will consist of side- lying hip abduction, hip external rotation (clamshell), and prone hip extension.
  2. Knee-focused exercise The knee-focused exercise regime will be based on previous studies and consist of supine straight leg raises, supine terminal knee extensions (from 10° flexion to full extension), and a mini squat (45° flexion) with the back supported against the wall (to reduce stabilizing requirements from the hip muscles).
  Interventions: Other: Traditional treatment

INTERVENTIONS:
Other: Core strengthening exercises — By core strengthening exercise, could be improved pain, balance, and function in patients with patellofemoral pain syndrome. In that case, this will not only improve their postural stability and neuromuscular control, but we believe it will improve their overall functional, performance, and quality of life. Currently, limited evidence exists about the effectiveness of core strengthening exercises on pain, function and dynamic balance in patellofemoral pain syndrome. By addressing core strengthening exercise, physical therapists can advise new treatment methods for patellofemoral pain syndrome (Chevidikunnan et al., 2016)
  Arms: Study group
Other: Traditional treatment — hip and knee-focused exercises

SUMMARY:
the goal of this interventional study is to Investigate the effect of core strengthening exercises on pain, strength, function, and balance in patients with PFPS.

DETAILED DESCRIPTION:
Purpose: Patellofemoral pain syndrome is a frequent musculoskeletal disorder, which can result from core muscles instability that can lead to pain, function and altered dynamic balance. The objective of this study is to assess the effect of core muscle strengthening on pain, function, strength and dynamic balance in patients with patellofemoral pain syndrome.

Subjects and Methods: Forty-four patients with age ranging from 18 to 35 years with patellofemoral pain syndrome will be divided into study (N=22) and control (N=22) groups. Both groups will be given 6 weeks of conventional physical therapy program and an additional core muscle strengthening for the study group. The tools are being used to assess the outcome are 1- Visual Analogue Scale,2- handheld dynamometer,3-AKPS 4- BIODEX Balance.

Hypotheses:

It will be hypothesized that:

1. There is no effect of core strengthening exercises on pain in treating PFPS.
2. There is no effect of core strengthening exercises on muscle strength in treating PFPS.
3. There is no effect of core strengthening exercises on function in treating PFPS.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of both genders with an age range of 18- 35 years old.
2. Gradual development of pain in the front of the knee lasting more than 12 weeks.
3. Patients with body mass index 18- 25 kg m2.
4. Pain is aggravated by at least 2 of the following activities: jumping, running, prolonged sitting, stair climbing, kneeling, and squatting.

   1. Positive patellar grinding test.
   2. Insidious onset of symptoms, unrelated to a traumatic damage.

Exclusion Criteria:

1. Traumatic patellar subluxation or dislocation.
2. A history of any of the following conditions: meniscal or other intra articular pathologic conditions; cruciate or collateral ligament involvement.
3. Any lower limb bony or congenital deformities.
4. Previous knee and hip joint surgeries.
5. Osteoarthritis in the ankle, knee, or hip joints.
6. Conditions that affect muscle strength such as diabetes mellitus or rheumatoid arthritis.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Estimated)
Dates: Start 2024-08-04 (Actual); Primary Completion 2025-01-15 (Estimated); Study Completion 2025-01-30 (Estimated)

PRIMARY OUTCOMES:
Pain | 6 weeks
  by Visual analog scale
knee function | 6 weeks
  by Anterior knee pain scale ( AKPS) ( Kujala )

SECONDARY OUTCOMES:
Muscle strength | 6 weeks
  By hand held dynamometer
Balance | 6 weeks
  By Biodex balance system

CONTACTS AND LOCATIONS:
Overall Officials: rana ibrahim ahmed, Bachelor Physical Therapy-MUST, Principal Investigator — Misr University for Science and Technology; Nasr Awad Abd Elkader, Assistant Professor, Study Chair — Physical Therapy for Musculoskeletal Disorders and its Surgeries Faculty of Physical Therapy Cairo University; Abdelgalil Allam Abdelgalil, Lecturer of Physical Therapy, Study Director — Physical Therapy for Musculoskeletal Disorders and its Surgeries Faculty of Physical Therapy Cairo University; Mohammed Safwat Hamza, Associate Professor, Study Director — Faculty of Medicine Misr University for Science and Technology
Locations (1):
- Cairo University, Giza, Egypt